CLINICAL TRIAL: NCT01970475
Title: A Randomized, Double-blind, Phase 3 Study of ABP 501 Efficacy and Safety Compared to Adalimumab in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: Efficacy and Safety Study of ABP 501 Compared to Adalimumab in Subjects With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120262; 2013-000525-31 (EudraCT Number)
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis; Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — ABP 501; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABP 501 (Experimental): Participants received ABP 501 40 mg subcutaneously on day 1 and every 2 weeks thereafter until week 22.
  Interventions: Biological: ABP 501
- Adalimumab (Active Comparator): Participants received adalimumab 40 mg subcutaneously on day 1 and every 2 weeks thereafter until week 22.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: ABP 501 — Solution for subcutaneous injection in pre-filled syringe
  Other Names: AMJEVITA™; Adalimumab-atto
  Arms: ABP 501
Biological: Adalimumab — Solution for subcutaneous injection in pre-filled syringe
  Other Names: HUMIRA®
  Arms: Adalimumab

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of ABP 501 against adalimumab (HUMIRA®) in adults with moderate to severe rheumatoid arthritis (RA) who have an inadequate response to methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 and ≤ 80 years old
2. Subjects must be diagnosed with rheumatoid arthritis for at least 3 months before baseline
3. Active RA defined as ≥ 6 swollen joints and ≥ 6 tender joints at screening and baseline
4. Subjects must be taking MTX for ≥ 12 consecutive weeks and on a stable dose of 7.5 to 25 mg/week for > 8 weeks prior to receiving the study drug and be willing to remain on stable dose throughout the study
5. Subject has no known history of active tuberculosis

Exclusion Criteria:

1. Class IV RA, Felty's syndrome or history of prosthetic or native joint infection
2. Major chronic inflammatory disease or connective tissue disease other than RA, with the exception of secondary Sjögren's syndrome
3. Prior use of 2 or more biologic therapies for RA
4. Previous receipt of HUMIRA® (adalimumab) or a biosimilar of adalimumab
5. Ongoing use of prohibited treatments

Other Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (5):
  - Research Site, Victorville, California
  - Research Site, Jupiter, Florida
  - Research Site, Sandy Springs, Georgia
  - Research Site, Lansing, Michigan
  - Research Site, Middleburg Heights, Ohio
- Research Site, Winnipeg, Manitoba, Canada
- Research Site, Hattingen, North Rhine-Westphalia, Germany
- United Kingdom (4):
  - Research Site, Barnsley, England
  - Research Site, North Shields, England
  - Research Site, Suffolk, England
  - Research Site, Cardiff, Wales

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Cohen S, Genovese MC, Choy E, Perez-Ruiz F, Matsumoto A, Pavelka K, Pablos JL, Rizzo W, Hrycaj P, Zhang N, Shergy W, Kaur P. Efficacy and safety of the biosimilar ABP 501 compared with adalimumab in patients with moderate to severe rheumatoid arthritis: a randomised, double-blind, phase III equivalence study. Ann Rheum Dis. 2017 Oct;76(10):1679-1687. doi: 10.1136/annrheumdis-2016-210459. Epub 2017 Jun 5. PMID 28584187
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 92 centers in 12 countries in Europe, North America and Latin America.
  The first participant enrolled on 24 October 2013 and the last participant enrolled on 26 May 2014.
Pre-assignment Details: Participants were randomized 1:1 to receive either ABP 501 or adalimumab at 40 mg every 2 weeks for 22 weeks. Randomization was stratified by geographic region and prior biologic use for rheumatoid arthritis (capped at 40% of the study population).
Period: Overall Study
Arm/Group | ABP 501 | Adalimumab
Started | 264 | 262
Completed | 243 | 251
Not Completed | 21 | 11
Not completed — Withdrawal by Subject | 11 | 6
Not completed — Adverse Event | 7 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (all randomized participants)
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP 501 | Adalimumab | Total
Number analyzed (Participants) | 264 | 262 | 526
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.88) | 56.3 (11.47) | 55.9 (11.67)
Age, Customized [Number; unit: participants]
  < 65 years | 205 | 197 | 402
  ≥ 65 years | 59 | 65 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 212 | 426
  Male | 50 | 50 | 100
Race/Ethnicity, Customized [Number; unit: participants]
  White | 251 | 249 | 500
  Black or African American | 9 | 12 | 21
  Asian | 3 | 0 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 1 | 2
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 33 | 25 | 58
  Not Hispanic or Latino | 230 | 236 | 466
  Not Allowed to Collect | 1 | 1 | 2
Geographic Region [Number; unit: participants]
  Eastern Europe | 169 | 168 | 337
  Western Europe | 22 | 20 | 42
  North America | 72 | 72 | 144
  Latin America | 1 | 2 | 3
Prior Biological Use for Rheumatoid Arthritis (RA) [Number; unit: participants]
  Yes | 71 | 74 | 145
  No | 193 | 188 | 381
Duration of RA [Mean (Standard Deviation); unit: years] | 9.41 (8.076) | 9.37 (8.047) | 9.39 (8.054)
Swollen Joint Count [Mean (Standard Deviation); unit: swollen joints] — Sixty-six joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination.
  swollen joints | 14.7 (9.05) | 14.1 (7.98) | 14.4 (8.53)
Tender Joint Count [Mean (Standard Deviation); unit: tender joints] — Sixty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination.
  tender joints | 24.3 (14.35) | 23.9 (13.49) | 24.1 (13.92)
Subject Global Health Assessment [Mean (Standard Deviation); unit: units on a scale] — The participant's overall assessment of their disease activity in the past week on a 0 to 10 horizontal scale. The left-hand extreme of the scale was described as "no RA activity at all" (symptom-free and no arthritis symptoms; score = 0) and the right-hand extreme as "worst RA activity imaginable" (maximum arthritis disease activity; score = 10).
  units on a scale | 6.5 (1.92) | 6.6 (1.86) | 6.5 (1.89)
Investigator Global Health Assessment [Mean (Standard Deviation); unit: units on a scale] — The Investigator's assessment of the participant's current disease activity on a 0 to 10 horizontal scale. The left-hand extreme of the scale was described as "no activity at all" (symptom-free and no arthritis symptoms; score = 0) and the right-hand extreme as "worst activity imaginable" (maximum arthritis disease activity; score = 10).
  units on a scale | 6.8 (1.29) | 6.7 (1.59) | 6.8 (1.45)
Subject's Assessment of Disease Related Pain [Mean (Standard Deviation); unit: units on a scale] — The participant's assessment of their current level of pain on a 100 mm horizontal visual analogue scale (VAS). The left-hand extreme of the line was described as "no pain at all" (score = 0) and the right-hand extreme as "worst pain imaginable" (score = 100).
  units on a scale | 58.3 (21.82) | 60.6 (22.37) | 59.5 (22.11)
Health Assessment Questionnaire-Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The HAQ-DI questionnaire asks participants to rate their level of difficulty on daily activities as well as their use of aids, devices, or help from another person for these activities and disabilities. Responses are scored from 0 indicating no difficulty to 3 indicating inability to perform a task in that area. The overall score is the average of each of the 8 category scores and ranges from 0 (no disability) to 3 (very severe, high-dependency disability).
  Data are available for 263 and 261 participants in each group respectively.
  units on a scale | 1.4819 (0.61715) | 1.4976 (0.64743) | 1.4897 (0.63186)
C-reactive Protein [Mean (Standard Deviation); unit: mg/L] | 13.881 (20.6870) | 14.678 (19.3848) | 14.278 (20.0338)
Disease Activity Score 28-C-Reactive Protein (DAS28-CRP) [Mean (Standard Deviation); unit: units on a scale] — The DAS28-CRP is a composite score to measure disease activity in patients with RA, derived from the following variables:
  * The number of swollen and tender joints (28-joint count);
  * C-reactive protein (CRP);
  * Patient's global assessment of disease activity assessed on a scale from 0 to 100 transformed from the result measured on a horizontal scale from 0 (no RA activity at all) to 10 (worst RA activity imaginable).
  DAS28-CRP scores range from approximately zero to ten. Higher scores indicate higher disease activity.
  Data are available for 264 and 261 participants in each group respectively.
  units on a scale | 5.66 (0.918) | 5.68 (0.911) | 5.67 (0.914)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response at Week 24
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 20% improvement in tender joint count;
  * ≥ 20% improvement in swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Physician's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-Reactive Protein level.
Time Frame: Baseline and Week 24
Population: The full analysis set (all randomized participants); missing values were imputed using the last observation carried forward (LOCF) method for participants with at least 1 postbaseline value.
Measure: Number; unit: percentage of participants
Arm/Group | ABP 501 | Adalimumab
Number analyzed (Participants) | 260 | 261
percentage of participants | 74.6 | 72.4
Statistical Analysis 1: Comparison: ABP 501 vs Adalimumab; The study hypothesis was that there were no clinically meaningful differences between ABP 501 and adalimumab in risk ratio (RR) of ACR20 at week 24; Test type: Non-Inferiority or Equivalence — The hypothesis was tested by comparing the 2-sided 90% confidence interval (CI) of the RR of ACR20 at week 24 between ABP 501 and adalimumab with an equivalence margin of (0.738, 1/0.738); Risk Ratio (RR) = 1.039, 90% CI 2-sided [0.954 to 1.133] — Based on a generalized linear model adjusted for geographic region and prior biological use for RA as covariates in the model

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28-C-reactive Protein (DAS28-CRP)
Description: The DAS28-CRP is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * C-reactive protein (CRP) level
  * Patient's global assessment of disease activity assessed on a score from 0 to 100 transformed from the result measured on a horizontal scale from 0 (no RA activity at all) to 10 (worst RA activity imaginable).
  The DAS28-CRP score ranges from approximately zero to ten. Higher DAS28-CRP scores indicate higher disease activity.
  A repeated measures analysis with the DAS28-CRP change from baseline as the response and the stratification variables, visit, treatment, treatment-by-visit interaction and the baseline DAS28-CRP measurement as predictors in the model was performed.
Time Frame: Baseline and weeks 2, 4, 8, 12, 18, and 24
Population: Full analysis set with available data at each time point
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP 501 | Adalimumab
Number analyzed (Participants) | 264 | 262
units on a scale
  Week 2 (n = 254, 252) | -1.01 (0.891) | -0.96 (0.890)
  Week 4 (n = 255, 254) | -1.45 (1.048) | -1.42 (0.979)
  Week 8 (n = 247, 255) | -1.79 (1.075) | -1.70 (1.093)
  Week 12 (n = 245, 250) | -2.04 (1.112) | -1.93 (1.171)
  Week 18 (n = 244, 250) | -2.30 (1.184) | -2.17 (1.189)
  Week 24 (n = 243, 250) | -2.32 (1.237) | -2.32 (1.209)

3. Secondary Outcome: Percentage of Participants With an ACR20 Response at Week 2 and Week 8
Description: as for outcome 1
Time Frame: Baseline, week 2 and week 8
Population: Full analysis set; LOCF imputation was used for participants with at least 1 postbaseline value (indicated by n).
Measure: Number; unit: percentage of participants
Arm/Group | ABP 501 | Adalimumab
Number analyzed (Participants) | 264 | 262
percentage of participants
  Week 2 (n = 254, 257) | 35.4 | 24.5
  Week 8 (n = 260, 261) | 63.5 | 62.5

4. Secondary Outcome: Percentage of Participants With an ACR50 Response at Week 24
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Physician's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-Reactive Protein level.
Time Frame: Baseline and week 24
Population: Full analysis set with available data at week 24
Measure: Number; unit: percentage of participants
Arm/Group | ABP 501 | Adalimumab
Number analyzed (Participants) | 244 | 252
percentage of participants | 49.2 | 52.0

5. Secondary Outcome: Percentage of Participants With an ACR70 Response at Week 24
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Physician's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-Reactive Protein level.
Time Frame: Baseline and Week 24
Population: Full analysis set with available data at week 24
Measure: Number; unit: percentage of participants
Arm/Group | ABP 501 | Adalimumab
Number analyzed (Participants) | 246 | 253
percentage of participants | 26.0 | 22.9

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 according to the following scale:
  1 = mild; 2 = moderate; 3 = severe; 4 = life-threatening; 5 = fatal. A treatment-related AE is defined as an event where the answer to the question "is there a reasonable possibility that the event may have been caused by the Investigational Medicinal Product" was yes.
  A serious adverse event is defined as an AE that meets at least 1 of the following serious criteria:
  * fatal
  * life threatening (places the subject at immediate risk of death)
  * requires inpatient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event.
Time Frame: From the time of first treatment up to 28 days following the last dose of study treatment; 26 weeks.
Population: The safety analysis set (all participants who received at least 1 dose of study drug)
Measure: Number; unit: participants
Arm/Group | ABP 501 | Adalimumab
Number analyzed (Participants) | 264 | 262
participants
  Any adverse event (AE) | 132 | 143
  Adverse event ≥ grade 3 | 9 | 17
  Treatment-related adverse event (TRAE) | 50 | 55
  Treatment-related adverse event ≥ grade 3 | 3 | 2
  Serious adverse event (SAE) | 10 | 13
  Treatment-related serious adverse event | 4 | 1
  AE leading to discontinuation of study drug | 5 | 2
  TRAE leading to discontinuation of study drug | 4 | 1
  AE leading to discontinuation from study | 7 | 2
  TRAE leading to discontinuation from study | 5 | 0

7. Secondary Outcome: Percentage of Participants Who Developed Antibodies to ABP 501 or Adalimumab
Description: Two validated assays were used to detect the presence of anti-drug antibodies. Samples were first tested in an electrochemiluminescence (ECL)-based bridging immunoassay to detect anti-drug antibodies (ADA) against ABP 501 and adalimumab (Binding Antibody Assay). Samples confirmed to be positive for binding antibodies were subsequently tested in a non-cell based bioassay to determine neutralizing activity against ABP 501 or adalimumab (Neutralizing Antibody Assay).
  Developing antibody incidence is defined as a negative or no antibody result at baseline and a positive antibody result at a post-baseline time point.
Time Frame: Up to week 26
Population: Participants with at least 1 evaluable antibody test result (to either ABP 501 or adalimumab)
Measure: Number; unit: percentage of participants
Arm/Group | ABP 501 | Adalimumab
Number analyzed (Participants) | 264 | 262
percentage of participants
  Developing Binding Antibody | 38.3 | 38.2
  Developing Neutralizing Antibody | 9.1 | 11.1

ADVERSE EVENTS:
Time Frame: From the time of first treatment but on or within 28 days following the last dose of study treatment; 26 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | ABP 501 | Adalimumab
Serious Adverse Events (participants affected / at risk) | 10/264 | 13/262
Other Adverse Events (participants affected / at risk) | 17/264 | 19/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 501 (N=264) | Adalimumab (N=262)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Corneal graft rejection (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Peritoneal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 501 (N=264) | Adalimumab (N=262)
Nasopharyngitis (Infections and infestations) | 17 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.